CLINICAL TRIAL: NCT00492739
Title: Induction and Maintenance of Immunity Against Varicella in Pediatric Orthotopic Liver Transplantation Recipients: a Retrospective and Prospective Nationwide Study in Switzerland
Brief Title: Immunity Against Varicella in Pediatric Orthotopic Liver Transplantation Recipients
Acronym: VZVinOLTx
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Klara M. Pósfay Barbe, Head of Pediatric Infectious Diseases, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VZVinOLTx
Record Dates: First submitted 2007-06-22; First posted 2007-06-27 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Liver Disease; Immunosuppression; Varicella
Keywords: Orthotopic liver transplantation; Pediatric; Immunosuppression; Varicella vaccine; B cell response; T cell response; Antibodies; Varicella; Chickenpox; transplantation
MeSH Terms: conditions — Liver Diseases; Chickenpox | interventions — Vaccination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Varicella vaccine (Other): 2-3 doses of Varicella vaccine to seronegative patients two months apart
  Interventions: Biological: Vaccination with VZV vaccine

INTERVENTIONS:
Biological: Vaccination with VZV vaccine — Varicella vaccination 2 doses 2 months apart.
  Other Names: Varilrix

SUMMARY:
Varicella is a vaccine-preventable disease, which can be severe in immunosuppressed children. Currently, the (live) vaccine is not recommended in pediatric orthotopic liver transplant recipients. Furthermore, protection due to naturally acquired immunity to VZV or post-immunization isn't well described in this population.The questions asked are:

* What is the influence of the immunosuppression required after orthotopic liver transplantation (OLT) on the maintenance of VZV-specific immunity elicited by wild-type varicella infection before OLT transplantation?
* What is the influence of the immunosuppression required after OLT on VZV-specific immunity elicited by varicella immunization before OLT transplantation?
* What is the influence of the residual immunosuppression at ≥ 12 months after OLT transplantation on the induction of VZV-specific B and T cell responses elicited by VZV vaccination after OLT transplantation?
* What is the influence of the residual immunosuppression at ≥ 12 months after OLT transplantation on the persistence / waning of B and T cell responses elicited by VZV vaccination?

DETAILED DESCRIPTION:
VZV vaccine given to pediatric liver transplant recipients at least one year after transplantation if tehy fulfill inclusion criteria and give informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Children either awaiting or recipients of a liver transplantation followed at the Children's Hospital of Geneva, Switzerland
* If vaccination offered: > 12 months of age

Exclusion Criteria:

* Known wild type varicella exposure within four weeks of the initial vaccine
* Immunoglobulins administered within the 5 months preceding the receipt of varicella vaccine.
* Antiviral agents administered during the preceding 4 weeks
* Febrile illness (>38.5°) in the 72 hours before vaccine administration
* Chronic aspirin therapy
* Any other live vaccinations within four weeks of receipt of varicella vaccine
* Female patients in childbearing age will have a pregnancy test at enrollment, and at the time of the second vaccine.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-06; Primary Completion 2022-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety of VZV vaccine in OLTx recipients | 2 years
  Antibody response measured after vacination with long-term f/u

SECONDARY OUTCOMES:
Efficacy of VZV vaccine in immunosuppressed OLTx recipients | 3 years
  Protection from disease monitored

CONTACTS AND LOCATIONS:
Overall Officials: Klara M Posfay-Barbe, MD, MS, Principal Investigator — University Hospitals of Geneva
Locations (1):
- Children's Hospital of Geneva (HUG), Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suresh S, Upton J, Green M, Pham-Huy A, Posfay-Barbe KM, Michaels MG, Top KA, Avitzur Y, Burton C, Chong PP, Danziger-Isakov L, Dipchand AI, Hebert D, Kumar D, Morris SK, Nalli N, Ng VL, Nicholas SK, Robinson JL, Solomon M, Tapiero B, Verma A, Walter JE, Allen UD. Live vaccines after pediatric solid organ transplant: Proceedings of a consensus meeting, 2018. Pediatr Transplant. 2019 Nov;23(7):e13571. doi: 10.1111/petr.13571. Epub 2019 Sep 9. PMID 31497926
- [Background] Verolet CM, Pittet LF, Wildhaber BE, McLin VA, Rodriguez M, Grillet S, Siegrist CA, Posfay-Barbe KM. Long-term Seroprotection of Varicella-zoster Immunization in Pediatric Liver Transplant Recipients. Transplantation. 2019 Nov;103(11):e355-e364. doi: 10.1097/TP.0000000000002866. PMID 31335765
- [Background] Posfay-Barbe KM, Pittet LF, Sottas C, Grillet S, Wildhaber BE, Rodriguez M, Kaiser L, Belli DC, McLin VA, Siegrist CA. Varicella-zoster immunization in pediatric liver transplant recipients: safe and immunogenic. Am J Transplant. 2012 Nov;12(11):2974-85. doi: 10.1111/j.1600-6143.2012.04273.x. Epub 2012 Sep 20. PMID 22994936